CLINICAL TRIAL: NCT03604068
Title: Protocol For The Randomized Controlled Trial Of Pulsed Short Wave Therapy In Cesarean Section
Brief Title: Pulsed Short Wave Therapy In Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioElectronics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO180401
Record Dates: First submitted 2018-06-05; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain
Keywords: Caesarean section
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Group (Active Comparator): Patients in this group will be treated with the currently used standard protocol for the control of post-operative pain as well as an active RecoveryRx Pulsed Short Wave Therapy device.
  Interventions: Device: RecoveryRx
- Control Group (Sham Comparator): Patients in this group will be treated with the currently used standard protocol for the control of post-operative pain as well as a sham RecoveryRx Pulsed Short Wave Therapy device.
  Interventions: Device: Sham RecoveryRx

INTERVENTIONS:
Device: RecoveryRx — A pulsed shortwave therapy medical device
  Other Names: pulsed shortwave therapy
  Arms: Active Group
Device: Sham RecoveryRx — A sham pulsed shortwave therapy medical device
  Other Names: Sham pulsed shortwave therapy
  Arms: Control Group

SUMMARY:
This clinical study is designed to assesses the benefit of adding pulsed shortwave therapy to the postoperative pain and recovery protocol following Cesarean section. Pulsed shortwave therapy is a safe adjunct pain therapy for acute and chronic pain.

DETAILED DESCRIPTION:
Pain is ranked highest among undesirable clinical outcomes associated with caesarean section therefore postoperative pain relief following a cesarean section is extremely important to optimize maternal and neonate well being. Multimodial analgesics are effective in reducing postoperative pain but analgesia is still not optimized. Opiate based analgesics are effective but having troubling side effects. Addition of non-drug pain therapies hold promise in improving postoperative recovery while potentially allowing for reduced use of drug based analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily
* Performed using spinal anesthesia
* ASA I (Normal healthy patients) and II (Patients with mild systemic disease) (as defined by the American Society of Anesthesiologists Physical Status Classification system)
* PARA 0000, 1, 2, 3 [i.e. First, Second, or Third C-Section)
* At term pregnancy (>38 weeks)
* BMI <35
* Age between 18 - 50 years

Exclusion Criteria:

* Longitudinal surgical incision
* Placental abnormalities noted
* Time of extraction of the fetus >10 min from cutaneous incision
* Blood loss during surgery of >800 ml
* Any of the conditions not considered in inclusion criteria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Medication Use | Data collected daily for 7 Days
  Quantify the use of analgesic medications during 7 days of postoperative recovery.

SECONDARY OUTCOMES:
Change in Visual Analogue Pain | Data collected for 7 Days
  The visual analog scale (VAS) has been used extensively for rating pain intensity in previous studies. Postoperative pain will be measured daily over a 7 day recovery period
Time to patient Patient Mobility | 2 Days
  The benefits of mobility outlined in current nursing textbooks indicate that "Early ambulation is the most significant general nursing measure to prevent postoperative complications". There the time in hours after the c-section operation when the patient becomes mobile(walking) will be used recorded.
Would Closure at Day 7, Wound Complications | 7 Days
  presence of edema, erythema,hematoma, and exudate from the surgical wound on the seventh postoperative day that could impair woundhealing process

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa Chaaban, MD, Principal Investigator — Haykal hospital
Locations (2):
- Lebanon (2):
  - Haykal hospital, Tripoli
  - New Mazloum Hospital, Tripoli

REFERENCES:
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021